CLINICAL TRIAL: NCT02295150
Title: Prospective, Pharmacokinetic Study for Determination of the Relationship Between Lean Body Weight and Anti-Xa Activity 4 Hours After Subcutaneous Injection of 5700 IU Nadroparin in Morbidly Obese Patients After Bariatric Surgery.
Brief Title: Prophylaxis of Venous Thromboembolism After Bariatric Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Principal Investigator, Frits Berends, Dr., Rijnstate Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Frax001; 2012-002816-19 (EudraCT Number)
Record Dates: First submitted 2014-11-11; First posted 2014-11-20 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Morbid Obesity; Thromboembolism; Bypass Complications
Keywords: Nadroparin; Anti-Xa activity
MeSH Terms: conditions — Obesity, Morbid; Thromboembolism | interventions — Nadroparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nadroparin (Experimental): patients above 140 kg will receive a dose of 2850 IU nadroparine pre-operatively, anti-Xa factor will be determined 3 days after nadroparin use. After surgery patients receive 5700 IU nadroparin (our standard treatment). Three days after surgery and 4 weeks after surgery anti-Xa factor will be measured again.
  Interventions: Drug: Nadroparin

INTERVENTIONS:
Drug: Nadroparin — Patients receive before surgery 3 days 2850 IU nadroparin. anti-Xa levels will be measured. After surgery they receive 5700 IU for 4 weeks as standard care in our hospital. 3 days and 4 weeks after surgery anti-Xa levels will be measured again.
  Other Names: Fraxiparin

SUMMARY:
This study is a prospective evaluation of the relationship between lean body weight and anti-Xa activity and 5700 International Units (IU) nadroparin 4 hours after subcutaneous administration in morbidly obese patients after bariatric surgery.

DETAILED DESCRIPTION:
There is no guideline for postoperative thromboembolic prevention in morbidly obese patients.

The investigators goal is to examine which dose of nadroparin is effective.

ELIGIBILITY:
Inclusion Criteria:

* Approval for Roux-en-Y gastric bypass
* Total body weight > 140 kg

Exclusion Criteria:

* Renal impairment (GFR < 30ml/min and/ or serum creatinin > 150 micromol/ml)
* Coagulation disorders
* Use of vitamin K antagonists (such as acenocoumarol) pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
anti-Xa activity 4 hours after subcutaneous administration of 5700 IU nadroparin | 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: F.J. Berends, MD, PhD, Principal Investigator — Rijnstate Hospital
Locations (1):
- Rijnstate Hospital, Arnhem, Wagnerlaan 55, Netherlands